CLINICAL TRIAL: NCT06753162
Title: Oral Health Perception Among 4,079 Women With Endometriosis: A Cohort Study
Brief Title: Oral Health and Endometriosis: A Cohort Study
Acronym: Oral-Endomet
Status: Completed | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Other Study IDs: endometriosis-oralhealt
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis
Keywords: endometriosis; Oral Health; Periodontitis; Gengivitis
MeSH Terms: conditions — Endometriosis; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A survey has been conducted thanks to a questionnaire composed of 45 questions. The study group was composed of 4079 women affected by endometriosis, recruited from dedicated communities present on the social network Facebook. The questionnaire investigated about: the endometriosis status, the kind of therapy, the presence of any sign and symptoms in the oral cavity, the presence of periodontal problems, the self-perception of the oral health status, the presence of other autoimmune diseases and oral hygiene and the eating habits, physical activity practiced, the life quality.

DETAILED DESCRIPTION:
The questions were structured thanks to the collaboration of expert health professionals: gynecologist, dentist, dental hygienist, physiotherapist, dietician, psychologist to obtain targeted information on endometriosis, on the type of therapy, on any signs and symptoms in the oral cavity (perception health status, presence of periodontal problems), to investigate oral hygiene and dietary habits, physical activity, quality of life, the presence of other immune-based diseases. In the final part of the questionnaire there was a section in which women were free to tell their stories.

ELIGIBILITY:
Inclusion Criteria:

* The only inclusion criterion was being at least 18 years old

Exclusion Criteria:

* • Pregnancy.

  * Administration of antibiotics in the last 15 days prior to entry into the study or indications for antibiotic prophylaxis.
  * Orthodontic Appliances.
  * Immunological diseases or use of drugs that can affect oral tissues (phenytoin, cyclosporine), nifedipine, chronic use of nonsteroidal anti-inflammatory drugs.
  * Refusal to participate in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women suffering from endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 4079 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Response Patterns Based on Multiple Correspondence Analysis Dimensions | 1 year
  To evaluate the possible correlations between endometriosis and the perception of periodontal disease, a score was created to summarize on a numerical scale the responses to survey questions describing the perception of oral cavity disorders. Multiple Correspondence Analysis (MCA) was used to explore relationships between responses. For the MCA, only questions with a p-value < 0.25 in the univariate analysis were included. The responses to the questions were labeled as "yes," "no," and "I don't know". In the case of question Q11, a grade was assigned to the responses as follows: "Idk" (I don't know), "Grd0" (Insufficient), "Grd1" (Average), "Grd2" (Good), "Grd3" (Very Good), and "Grd4" (Perfect).
Epidemiological Analysis | 1 year
  It was statistically evaluated whether the severity of endometriosis increased significantly with age.
Comparative Analysis of Oral Cavity Disorders Across Different Stages of Endometriosis | 1 year
  The correlation between general gum bleeding and the stage of the disease was statistically evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Saverio Capodiferro, Professor, Study Director — University of Bari Aldo Moro; Massimo Corsalini, Professor, Study Director — University of Bari Aldo Moro; Giuseppe D'Albis, Principal Investigator — University of Bari Aldo Moro; Agneta Maria Teresa, Principal Investigator — University of Bari Aldo Moro
Locations (1):
- University of Bari Aldo Moro, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided